CLINICAL TRIAL: NCT03929159
Title: Profile of miRNA Changes in Sepsis and Surgical Trauma
Brief Title: Correlating MicroRNA Changes With Sepsis Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0757; NCI-2019-00833 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0757 (Other: M D Anderson Cancer Center); R01GM122775 (NIH)
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (biospecimen collection): Patients undergo blood specimen collection at baseline (before surgery), the day after surgery, either the day of hospital discharge or the day of sepsis diagnosis, and 6 days after the baseline blood draw if still hospitalized.
  Interventions: Procedure: Biospecimen Collection
- Group B (biospecimen collection): Patients undergo blood specimen collection at baseline (day of sepsis diagnosis), the day after baseline, and on day 7 from baseline if still hospitalized.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood biospecimen collection

SUMMARY:
This trial studies how changes in microRNAs may correlate with sepsis outcomes. Sepsis is a type of severe infection of the blood stream, and its diagnosis may be obscured by many other conditions such as surgery, trauma, and cancer. MicroRNAs are biomarkers found in the blood and tissue. Blood samples may help correlate changes in microRNA expression to patient reactions to a sepsis infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine whether the cellular and viral micro ribonucleic acid (miRNA) changes in plasma and peripheral mononuclear blood cells (PMNCs) correlate with the diagnosis and outcome of sepsis.

SECONDARY OBJECTIVES:

I. To distinguish systemic inflammatory response syndrome (SIRS) without infection from sepsis and septic shock.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A: Patients undergo blood specimen collection at baseline (before surgery), the day after surgery, either the day of hospital discharge or the day of sepsis diagnosis, and 6 days after the baseline blood draw if still hospitalized.

GROUP B: Patients undergo blood specimen collection at baseline (day of sepsis diagnosis), the day after baseline, and on day 7 from baseline if still hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Electively scheduled for surgical operation that require general anesthesia and expected duration of hospitalization of longer than one day (for patients in Perioperative Evaluation & Management [POEM]) or high clinical suspicion of sepsis by the emergency physician (for patients in emergency center)
* Ability to give informed consent. If the patient is incapacitated and unable to give informed consent, the next-of-kin or a person who has the power of attorney must be present for informed consent.
* For patients in the emergency center only, two or more of the following SIRS criteria:

  * Leukocytes > 12,000/mm^3 or < 4,000/mm^3 or > 10% immature (band) forms, provided that no filgrastim or pegfilgrastim was administered within 30 days and no leukemia
  * Heart rate > 90 beats/minute (min)
  * Respiratory rate > 20 breaths/min or partial pressure of carbon dioxide (CO2) < 32 mmHg
  * Oral temperature > 38 degrees Celsius (C) or < 36 degrees C or axillary temperature > 37 degrees C or < 35 degrees C

Exclusion Criteria:

* Inability to give informed consent or a person who has power of attorney for medical decision is not available
* Being moribund (for patients in emergency center) or cancellation of surgery (for patients in POEM)
* Active "Do Not Resuscitate" or "Do Not Intubate" order

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients electively scheduled for surgical operation requiring anesthesia and hospitalization of longer than 1 day, or patients with high clinical suspicion of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cellular and viral micro ribonucleic acids (miRNAs) | Baseline up to day 1
  For each of the cellular and viral miRNAs, samples from patients with sepsis versus (vs.) patients with systemic inflammatory response syndrome (SIRS) without sepsis vs. patients presenting for pre-op evaluation (reference group without SIRS or sepsis) will be compared by one-way analysis of variance. Will compare the miRNA expression intergroup differences.
7-day mortality rate | Baseline up to day 7
  Will be correlated with miRNA changes. Will compare the changes of the miRNAs from baseline to day 1 between the patients who were still alive 7 days after diagnosis of sepsis and those who died within 7 days of sepsis diagnosis.

SECONDARY OUTCOMES:
T and B cells immune phenotypes | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Ching J Yeung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org